CLINICAL TRIAL: NCT01136720
Title: Clinical Trial to Evaluate the Safety and Clinical Utility of18F-FDG Produced by the Molecular Imaging and Research Centre of Nova Scotia
Brief Title: Clinical Trial to Evaluate the Safety and Clinical Utility of 18F-FDG Produced by the Molecular Imaging and Research Centre of Nova Scotia
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-035
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2022-10

CONDITIONS: 18FDG

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients injected with the Halifax produced 18-FDG

SUMMARY:
18F-FDG produced in the MIRC NS has a similar safety profile to the same compound utilized elsewhere in that no significant adverse events will occur during observation of the patients for 2 1/2 hours post injection of the tracer. It is also hypothesized that as this FDG produced by similar methodology and its quality assurance assessed as in another jurisdictions will have similar performance parameters in patients with focal lung pathology to that previously determined.

DETAILED DESCRIPTION:
Positron Emission Tomography (PET) utilizing 18F-FDG is a nuclear medicine imaging technique evaluating glucose related metabolic processes providing information not obtainable from anatomic imaging . 18F-FDG PET scanning is used clinically in most developed countries and Canadian jurisdictions primarily in oncology patients and also in assessing myocardial viability and some neurological conditions.

The functional information obtained from 18F-FDG PET has been demonstrated to have a significant impact on patient management in oncology.1 It is used to provide accurate pre-treatment staging, aid in planning of therapy, monitoring response to therapy, restaging, providing assessment of recurrence after curative therapy and in radiation treatment planning.

Patients with severe ischemic heart disease and secondary myocardial dysfunction pose difficult management decisions in terms of surgical vs. medical management. Assessment of viable myocardium is integral in this decision and 18F-FDG PET has been shown one of the most effective non-invasive methods in this evaluation.

18F-FDG PET has been shown very effective in neurology differentiating dementia types and in patients with epilepsy in whom surgical treatment is being considered.

The Capital District Health Authority (CDHA) PET/CT program has operated since June, 2008 and to date has examined over 2000 patients utilizing Health Canada approved 18F-FDG produced by Pharmalogic in Montreal. A significant component of the PET Program infrastructure in Nova Scotia is the Medical Imaging and Research Centre (MIRC NS) including a GMP grade radiopharmaceutical production lab and cyclotron. This CTA will allow evaluation of 18F-FDG produced at the MIRC-NS in a similar case load to prove its clinical utility and safety.

ELIGIBILITY:
Oncology

* Diagnosis to determine if a suspicious lesion is cancer
* Staging of confirmed cancer
* Evaluation of treatment response
* Follow up for cancer with high risk of recurrence
* Restaging following therapy
* Diagnosis of an unknown primary
* Assessment of potential paraneoplastic syndrome
* Radiation therapy planning

Neurology

18F-FDG PET will be used for evaluation of patients with

* Dementia, for differential diagnosis and prognosis
* Mild cognitive impairment, for suspected dementia
* Epilepsy, for localization of a seizure focus

Cardiology

• 18F-FDG PET in the evaluation of patients with ischemic heart disease and severely compromised myocardial function to aid in the evaluation of the appropriateness of revascularization.

General inclusion criteria:

* Diabetic patients are admissible, but will require proper control of their glucose levels (below 14) if possible prior to the scan.
* Receipt of an acceptably completed PET/CT scan requisition will be necessary.
* Patients will be able to tolerate the physical and logistic requirements of completing a PET scan including weight below 450lb and not claustrophobic to the extent that they can't tolerate being in the scanner gantry

EXCLUSION CRITERIA

* Pregnant women; if there is any possibility of pregnancy, a blood HCG level will be obtained
* Patients unwilling or unable to stop breast feeding for 24 hours
* Patients or guardians unwilling or unable to provide informed consent
* Patients who are medically unstable
* Patients who exceed the safe weight limit of the PET/CT bed or who cannot fit through the PET/CT gantry

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The recruited subjects will be patients referred by medical and surgical specialists involved in cancer management dementia epilepsy and cardiology
Sampling Method: Non-Probability Sample
Enrollment: 9463 (Actual)
Dates: Start 2010-06-19 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Ensure the Safety profile of the Halifax produced FDG is similar to litature based findings | 3 hours post injection
  The safety profile of the radiopharmaceutical will be monitored for adverse affects during the time in the department following injection. The technologists will inquire and note any potential signs or symptoms of adverse reactions. At the conclusion of the PET Centre visit, the patient will fill out a questionnaire assessing any potential adverse effects

SECONDARY OUTCOMES:
To effectively demonstrate diagnostic performance of the Halifax produced FDS in patients with focal lung pathology mirroring that previously published | 6 months
  The clinical efficacy will be analyzed in the patients with focal lung pathology. The clinical course of these patients will be followed to determine the true nature of these focal lesions with the gold standard being pathologic evaluation from either surgical procedure or biopsy results. In patients whom pathology is not made available, assessment of the lesion nature will be determined by other clinical indicators in consultation with the managing physicians opinion based upon these factors and the patient's clinical course.

CONTACTS AND LOCATIONS:
Locations (1):
- CapitalDHACanada, Halifax, Nova Scotia, Canada